CLINICAL TRIAL: NCT06496971
Title: A Prospective, Randomized, Standard of Care Controlled, Parallel, Open-Label, Multicenter Pivotal Study to Evaluate the Efficacy and Safety of Avastin® in Combination With NaviFUS System Compared With Avastin® Alone for the Treatment of Recurrent Glioblastoma Multiforme (rGBM)
Brief Title: A Prospective Pivotal Study to Evaluate the Efficacy and Safety of Avastin® Bevacizumab (BEV) With or Without Microbubble-mediated Focused Ultrasound (FUS-MB) Using NaviFUS System in Recurrent Glioblastoma Multiforme Patients
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: NaviFUS Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: NF-2023-01
Record Dates: First submitted 2024-07-01; First posted 2024-07-11 (Actual); Last update posted 2024-11-14 (Actual); Status verified 2024-11

CONDITIONS: Glioblastoma Multiforme; Glioblastoma; Glioblastoma Multiforme, Adult; Glioma; Brain Tumor; Brain Tumor, Recurrent; Neoplasms; Neoplasms, Nerve Tissue
Keywords: NaviFUS System; Blood-Brain Barrier Opening; Focused Ultrasound; FUS; Low-Intensity Focused Ultrasound; LIFU; Bevacizumab; BEV; Avastin
MeSH Terms: conditions — Glioblastoma; Glioma; Brain Neoplasms; Neoplasms; Neoplasms, Nerve Tissue | interventions — Bevacizumab; Microbubbles; contrast agent BR1

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Evaluators for radiological response assessment will be blinded to the patient's assigned treatment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard of care (SoC) BEV alone (Active Comparator): SoC group will follow the standard operating procedures of BEV (10 mg/kg intravenous (IV) infusion over 30-90 minutes, following the instructions in the drug package insert).
  Interventions: Drug: Bevacizumab
- Microbubble-mediated FUS treatment with BEV (FUS-MB+BEV) (Experimental): FUS-MB+BEV group will follow the standard operating procedures of BEV (10 mg/kg intravenous (IV) infusion over 30-90 minutes, following the instructions in the drug package insert). After at least 30 minutes, patients will be administered microbubbles (MB) (SonoVue® ) at a dose of 0.1 mL/kg, along with optimal ultrasound exposure doses determined by the acoustic emission feedback FUS power control algorithm of the NaviFUS System.
  Interventions: Drug: Bevacizumab; Drug: Microbubble; Device: Low-Intensity Focused Ultrasound

INTERVENTIONS:
Drug: Bevacizumab — An anti-angiogenic agent to block tumor growth
  Other Names: Avastin
Drug: Microbubble — Open the Blood-Brain Barrier (BBB) using focused ultrasound and microbubble
  Other Names: SonoVue
  Arms: Microbubble-mediated FUS treatment with BEV (FUS-MB+BEV)
Device: Low-Intensity Focused Ultrasound — Open the Blood-Brain Barrier (BBB) using focused ultrasound and microbubble
  Other Names: NaviFUS System
  Arms: Microbubble-mediated FUS treatment with BEV (FUS-MB+BEV)

SUMMARY:
This will be a prospective, randomized, standard of care (SoC) controlled, parallel, open-label, multicenter pivotal study to investigate the efficacy and safety of Bevacizumab (BEV) in combination with or without microbubble (MB)-mediated FUS in patients with recurrent GBM. BEV represents the physician's best choice for the standard of care in rGBM after previous treatment with surgery (if appropriate), standard radiotherapy with temozolomide chemotherapy, and with adjuvant temozolomide.

DETAILED DESCRIPTION:
The study aims to compare the efficacy of combining Bevacizumab with NaviFUS System relative to Bevacizumab alone in patients with rGBM who have previously undergone radiotherapy and temozolomide chemotherapy.

Any patient with a histological diagnosis of GBM who meets all of the specific eligibility criteria may participate in this study by signing informed consent in person or through their legal representative. Eligible patients will undergo a 2-week baseline observation screening period.

Up to 32 evaluable patients will be recruited in this study. Eligible patients will be randomized in a 1:1 ratio, with one group receiving the standard of care (SoC) BEV alone and the other group receiving treatment with microbubble-mediated FUS treatment in addition to BEV (FUS-MB+BEV).

Eligible patients who assigned to the SoC group will follow the standard operating procedures of BEV (10 mg/kg intravenous (IV) infusion over 30-90 minutes). On the other hand, eligible patients assigned to treatment group will initially receive the same BEV schedule. After at least 30 minutes, patients will be administered microbubbles (MB) (SonoVue® ) at a dose of 0.1 mL/kg, along with optimal ultrasound exposure doses determined by the acoustic emission feedback FUS power control algorithm of the NaviFUS System. The treatment will be administered every 2 weeks up to 34 weeks or until evidence of progression disease (PD), intolerable toxicity precluding further treatment, non- compliance with study follow-up, or withdrawal of consent, whichever occurs first.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female patients ≥ 18 years of age at the time of study enrollment.
2. Body mass index (BMI) ≥ 17 kg/m2.
3. Patients diagnosed with glioblastoma must have unequivocal evidence of recurrence, as determined by contrast-enhanced magnetic resonance imaging (CE-MRI), following prior radiotherapy and temozolomide chemotherapy.
4. Patients may have undergone surgery for recurrence. The patients should have completed surgery and adequately recovered prior to the time of study enrollment.
5. Patients must have radiographic evidence of either at least an 80% resection of enhancing tumor following recurrence or a maximal measurable residual tumor ≤ 20 cm3.
6. If patients are receiving corticosteroids, they must have been on a stable or decreasing dose of corticosteroids for at least 1 week prior to the planned first treatment.
7. At the time of study enrollment, the minimum interval since the last event:

   * 4 weeks out from invasive procedures (e.g., open biopsy, surgical resection, significant traumatic injury, or any other major surgery involving entry into a body cavity) and the patient must have recovered from the effects of surgery
   * 1 week out from minor surgical procedures or core biopsies
8. Patients must have recovered from the toxic effects of prior therapy at the time of study enrollment as follows:

   * 4 weeks out from any investigational drug or device
   * 4 weeks out from chemotherapy
   * 6 weeks since the completion of a nitrosourea-containing chemotherapy regimen (e.g., Carmustine (BCNU))
   * 12 weeks out from completion of radiotherapy
9. Patients should have a life expectancy ≥ 12 weeks.
10. Patients must have Karnofsky Performance Status (KPS) ≥ 70.
11. Adequate hematopoietic, renal, hepatic, and coagulation function, defined as:

    * Hemoglobin ≥ 10 g/dL
    * Platelets ≥ 100,000/mm3
    * Neutrophils ≥ 1,500/mm3
    * Serum creatinine ≤ 1.5 × upper limit of normal (ULN)
    * Urine protein creatinine ratio (UPCR) < 1 or urine dipstick for proteinuria ≤ 2+
    * Alanine aminotransferase (ALT) < 3 × ULN
    * Aspartate aminotransferase (AST) < 3 × ULN
    * Total bilirubin (TBL) < 2 × ULN
    * Prothrombin time ≤ 1.5 x ULN
    * International Normalized Ratio (INR) < 1.5 These tests must be conducted within 2 weeks prior to the planned first treatment.
12. The central of FUS exposure region is located with a minimum distance of at least 30 mm beneath the skull bone.
13. Females of childbearing potential must have a negative pregnancy test documented within 2 weeks prior to first treatment. Females of childbearing potential and male patients with partners of childbearing potential must agree to adhere to an acceptable method of contraception (as outlined below) from prior to the first study treatment until at least 6 months after the completion of last treatment. Standard acceptable methods of contraception include the use of highly effective methods such as hormonal contraception, diaphragm, cervical cap, vaginal sponge, condom, spermicide, vasectomy, intrauterine device, or abstinence from sexual activity.
14. Patients are able and willing to have peripheral intravenous (IV) line placement of Bevacizumab and are able to have hair shaved (either whole head or in the region where the coupling membrane will touch) prior to FUS treatment if assigned to treatment group.
15. Patients or their legal representatives are able to provide written informed consent for participation in the trial and patients are willing to comply the procedures (i.e., study-related assessments), instructions, and restrictions outlined in this study in the duration of the study. Informed consent should also be given for biological materials and diagnostic imaging to be stored and used for future research on brain tumors.

Exclusion Criteria:

1. Patients who have radiographic evidence of multifocal enhancing tumors.
2. Patients who have undergone previous treatment with anti-angiogenic therapy, including Bevacizumab, or other VEGF inhibitors or VEGF-receptor signaling inhibitors.
3. Patients who have previously received Carmustine wafers implantation during re-operation.
4. Patients who have previously received or are currently undergoing tumor treating fields (TTF) treatment.
5. Uncontrolled or significant cardiovascular disease, including any of the following:

   * New York Heart Association (NYHA) Grade II or above congestive heart failure (CHF) within 12 months prior to study enrollment
   * Unstable angina pectoris
   * Medical history of myocardial infarction within 6 months prior to study enrollment
   * Cardiac shunt
6. Stroke (except for transient ischemic attack; TIA) within 6 months prior to study enrollment.
7. Patients with implanted electronic device, for example, implanted cardioverter-defibrillator (ICD), cardiac pacemaker, permanent medication pumps, cochlear implants, responsive neurostimulator (RNS), deep brain stimulation (DBS), or other electronic devices implanted in the brain. Patients with contraindications for MRI as judged by Investigator, including non-MRI compatible metallic implant(s).
8. Patients with inadequately controlled hypertension, defined as systolic blood pressure > 150 mmHg and/or diastolic blood pressure > 100 mmHg while on medication, within 2 weeks prior to first treatment.
9. Patients with evidence of any thrombotic or hemorrhagic events, including but not limited to:

   * Inherited bleeding diathesis or significant coagulopathy with the risk of bleeding (i.e., in the absence of therapeutic anticoagulation).
   * History of pulmonary haemorrhage/haemoptysis ≥ grade 2 according to the CTCAE version 5.0 criteria within 1 month prior to study enrollment
   * Arterial or venous thrombosis (e.g., pulmonary embolism) within 3 months prior to study enrollment
10. Patients with unstable pulmonary disease or chronic obstructive pulmonary disease (COPD) exacerbation or other respiratory illness requiring hospitalization or precluding study therapy at the time of study enrollment.
11. Patients who have psychiatric illness/social situations that would limit compliance with study requirements.
12. Known HIV-positive patient, however, that HIV testing is not required for entry into this study.
13. Acute bacterial or fungal infection requiring intravenous antibiotics at the time of study enrollment.
14. History or evidence of active gastroduodenal ulcer, gastrointestinal perforations/fistula, or intra-abdominal abscess within 6 months prior to study enrollment.
15. Receiving anticoagulant (e.g., warfarin or LMW heparin) or antiplatelet (e.g., aspirin) therapy within 1 week prior to beginning treatment.
16. Known sensitivity/allergy to Magnetic Resonance Imaging (MRI) contrast agents, Computer Tomography (CT) contrast agents, SonoVue®, Bevacizumab, or any of their components.
17. Pregnant (positive pregnancy test) or breast-feeding women.
18. Use of any recreational drugs or history of drug addiction.
19. Other severe concurrent and/or uncontrolled concomitant medical conditions (e.g., active or uncontrolled infection, uncontrolled epilepsy, uncontrolled diabetes) that could cause unacceptable safety risks or compromise compliance with the protocol.
20. Any other condition that, in the Investigator's discretion, might increase the risk to the patients or compromise the evaluation of the clinical trial endpoints.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Estimated)
Dates: Start 2024-11-08 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-03-31 (Estimated)

PRIMARY OUTCOMES:
6-month progression-free survival (PFS-6) of Bevacizumab (BEV) with or without microbubble-mediated focused ultrasound (FUS-MB) using NaviFUS System | Up to 6 months
  PFS-6 will be estimated the proportion of patients who remain progression-free at the 6-month time point, based on Response Assessment in Neuro-Oncology (RANO) Criteria, from the time of randomization.

SECONDARY OUTCOMES:
12-month progression-free survival (PFS-12) | Up to 12 months
  PFS-12 will be estimated the proportion of patients who remain progression-free at the 12-month time point, based on Response Assessment in Neuro-Oncology (RANO) Criteria, from the time of randomization.
Progression-free survival time (PFS) | Up to 62 weeks
  PFS is defined as the time from the date of randomization to the earliest date of the first objective documentation of radiographic progression disease based on RANO Criteria, death, or last known follow-up due to any cause whichever occurs first. PFS will be followed continuously till the End-of-Study.
One- and Two-year survival rates | Up to 12 and 24 months
  One- and Two-year survival rates will be estimated the proportion of patients who remain alive at the one-year and two-year time points from the time of randomization.
Overall survival (OS) | Up to 36 months
  OS is defined as the time from the date of randomization to the earliest date of death or last known follow-up due to any cause whichever occurs first. OS will be followed continuously while subjects are on study and the survival follow-up phase of the study.
Objective response rate (ORR) | Up to 62 weeks
  ORR is defined as the proportion of patients who achieved a best overall response of complete response (CR) or partial response (PR) based on a combination of imaging and clinical features as assessed by the RANO Criteria.
Clinical benefit rate (CBR) | Up to 62 weeks
  CBR is defined as the proportion of patients who achieved an overall response of CR, PR, or stable disease (SD) based on a combination of imaging and clinical features as assessed by the RANO Criteria.
Local disease control on the MRI Images | Up to 62 weeks
  Local disease control is defined as the proportion of patients who achieved a CR, PR, or SD within the planning target tumor lesion, as assessed by the RANO Criteria. Progressive disease (PD) is defined as the presence of at least two sequential CE-MRI scans, separated by a ≥ 4 weeks interval, exhibiting local tumor progression at the treatment site, with distant recurrence or new lesion(s) not included in the assessment. The target tumor lesion on the MRI images will be assessed at baseline and throughout treatment period.
Corticosteroid consumption | Up to 62 weeks
  Corticosteroid consumption will be assessed at baseline and throughout treatment period. The mean corticosteroid dosage prior to study treatment will be considered as the patient's baseline. The changes in corticosteroids during treatment will be compared to baseline.
Severity and frequency of treatment-related adverse events (AEs) | Up to 62 weeks
  Documented and reported severity and frequency of AEs and/or SAEs will be assessed and classified based on National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) version 5.0.
Karnofsky performance status (KPS) | Up to 62 weeks
  The KPS score is rated on a scale of 0 to 100, where 0 represents death, and 100 represents normalcy without complaints or evidence of disease. A higher score indicates the patient is better able to perform daily activities.
Mini-Mental State Examination (MMSE) | Up to 62 weeks
  The MMSE is an 11-question measure that assesses multiple aspects of cognitive function. The maximum score is 30, with a higher score indicating less cognitive impairment.

CONTACTS AND LOCATIONS:
Locations (2):
- Taiwan (2):
  - National Taiwan University Hospital, Taipei
  - Linkou Chang Gung Memorial Hospital, Taoyuan District

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Liu HL, Hua MY, Chen PY, Chu PC, Pan CH, Yang HW, Huang CY, Wang JJ, Yen TC, Wei KC. Blood-brain barrier disruption with focused ultrasound enhances delivery of chemotherapeutic drugs for glioblastoma treatment. Radiology. 2010 May;255(2):415-25. doi: 10.1148/radiol.10090699. PMID 20413754
- [Background] Wei KC, Chu PC, Wang HY, Huang CY, Chen PY, Tsai HC, Lu YJ, Lee PY, Tseng IC, Feng LY, Hsu PW, Yen TC, Liu HL. Focused ultrasound-induced blood-brain barrier opening to enhance temozolomide delivery for glioblastoma treatment: a preclinical study. PLoS One. 2013;8(3):e58995. doi: 10.1371/journal.pone.0058995. Epub 2013 Mar 19. PMID 23527068
- [Background] Liu HL, Hsu PH, Lin CY, Huang CW, Chai WY, Chu PC, Huang CY, Chen PY, Yang LY, Kuo JS, Wei KC. Focused Ultrasound Enhances Central Nervous System Delivery of Bevacizumab for Malignant Glioma Treatment. Radiology. 2016 Oct;281(1):99-108. doi: 10.1148/radiol.2016152444. Epub 2016 May 18. PMID 27192459
- [Background] Chen KT, Lin YJ, Chai WY, Lin CJ, Chen PY, Huang CY, Kuo JS, Liu HL, Wei KC. Neuronavigation-guided focused ultrasound (NaviFUS) for transcranial blood-brain barrier opening in recurrent glioblastoma patients: clinical trial protocol. Ann Transl Med. 2020 Jun;8(11):673. doi: 10.21037/atm-20-344. PMID 32617293
- [Background] Chen KT, Chai WY, Lin YJ, Lin CJ, Chen PY, Tsai HC, Huang CY, Kuo JS, Liu HL, Wei KC. Neuronavigation-guided focused ultrasound for transcranial blood-brain barrier opening and immunostimulation in brain tumors. Sci Adv. 2021 Feb 5;7(6):eabd0772. doi: 10.1126/sciadv.abd0772. Print 2021 Feb. PMID 33547073
- See also: Related Info — http://classic.clinicaltrials.gov/ct2/show/NCT04446416